CLINICAL TRIAL: NCT03534115
Title: NAC Prevents Side-Effects of Teeth Bleaching
Brief Title: NAC Prevents Toxicity of Teeth Bleaching
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Anahid Jewett, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-001368
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Removal of Toxicity From Dental Bleaching
Keywords: bleaching, toxicity, NAC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: the investigators, clinical staff and patients were blinded. The main solution containing NAC or the placebo was marked by A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo was prepared by using the same solution containing buffers that were used in the preparation of NAC solution, except it did not contain NAC
  Interventions: Dietary Supplement: Placebo
- Experimental Arm (Experimental): solution containing NAC with buffers
  Interventions: Dietary Supplement: NAC

INTERVENTIONS:
Dietary Supplement: NAC — solution containing NAC
  Arms: Experimental Arm
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Dental bleaching is a simple procedure for aesthetic restoration of vital and non-vital discolored teeth. Nevertheless, a number of studies conducted previously demonstrated the risk of tissue damage from contact of these agents with the oral mucosa along with their possible genotoxic potential after exposure to oral mucosa. Hence the aim of this study is to conduct a human clinical trial to incorporate the chemoprotectant N-acetyl cysteine (NAC) in the procedure of bleaching which could safely be used to eliminate the toxicity of bleaching materials leaving their esthetic benefits intact. 30-40 human subjects will be recruited and bleaching will be done at the UCLA School of Dentistry dental clinic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be self reported as healthy individuals with no significant medical issues.

Exclusion Criteria:

* Self-report of present medical history (determined by the primary care doctors) of donors for:
* Pregnancy
* HIV-seropositivity and AIDS because the study is designed to evaluate the effect of NAC in general population with no underlying immunological deficiencies or general pathologies which may result in confounding effect in the outcome. Since this is a small study we are limiting the procedure to healthy individuals with no known underlying pathologies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
inhibition of pain | 3 weeks
  Patients self report of pain on a 0-10 pain scale with 10 being the highest for mean pain levels and 0-5 pain scale with 5 being the highest for resting pain levels.

SECONDARY OUTCOMES:
white lesion in gingiva | 3 weeks
  number and extend of white lesions in gingiva

IPD SHARING:
Plan to Share IPD: No